CLINICAL TRIAL: NCT05621668
Title: A First-In-Human Phase 1 Trial of T-Cell Membrane-Anchored Tumor Targeted Il12 (Attil12)- T-Cell Therapy in Subjects With Advanced/Metastatic Soft Tissue and Bone Sarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0619; NCI-2022-09675 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Soft Tissue Sarcoma; Bone Sarcoma
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose Findings (MTD) (Experimental): The dose of attIL2-T cell therapy the participants will receive will depend on when the participants joined this study. The first group of participants will receive the lowest dose level of attIL2-T cell therapy.
  Interventions: Drug: Cyclophosphamide; Drug: attIL2-T cells
- Part B: Osteosarcoma Dose Expansion (Experimental): Participants will receive attIL2-T cell therapy at the recommended dose that was found in Phase 1.
  Interventions: Drug: Cyclophosphamide; Drug: attIL2-T cells

INTERVENTIONS:
Drug: Cyclophosphamide — Given by IV (vein)
  Other Names: Cytoxan®; Neosar®
Drug: attIL2-T cells — Given by IV (vein)

SUMMARY:
To find a recommended dose of attIL2-T cell therapy that can be given to patients with soft tissue or bone sarcomas and to see if it can help to control the disease.

DETAILED DESCRIPTION:
Primary Objective:

1. Part A. Determine the safety, maximum tolerated dose and/or recommended phase 2 dose of adoptively transferred T cell membrane-anchored tumor targeted IL12 (attIL12)-T cells in combination with cyclophosphamide in patients with advanced/metastatic soft tissue or bone sarcomas
2. Part B. Characterize the safety and tolerability and assess preliminary efficacy of attIL12-armed T cells in combination with cyclophosphamide by evaluating the 4-month disease control rate (DCR4 months) in patients with recurrent unresectable osteosarcoma

Secondary Objectives:

1. Evaluate the anti-tumor efficacy achieved following adoptive transfer of T cellmembrane-anchored tumor targeted IL12 (attIL12)-T cells in combination with cyclophosphamide in patients with advanced/metastatic soft tissue or bone sarcomas

Exploratory Objectives:

1. Characterize the immune response following adoptive transfer of T cell membrane-anchored tumor targeted IL12 (attIL12)-T cells in paired in pre-treatment and on-treatment tumor specimens and peripheral blood samples
2. Assess FoxP3/CD33/CD8/IFNg expression in pre-treatment and on-treatment tumor specimens and correlate with clinical benefit/anti-tumor response
3. Determine changes in cell surface vimentin (CSV)-positive circulating tumor cells (CTCs) in peripheral blood before and after adoptive transfer of T cell membrane-anchored tumor targeted IL12 (attIL12)-T cells and correlate with clinical benefit/anti-tumor response

ELIGIBILITY:
Inclusion criteria:

1. Age .12 years old
2. Histologically-confirmed locally advanced or metastatic soft tissue or bone sarcoma
3. Osteosarcoma expansion cohort: histologically confirmed unresectable recurrent/metastatic osteosarcoma
4. Evaluable disease.
5. Patients must have received at least 1 prior line of systemic therapy for the treatment of sarcoma, unless no standard therapy exists for a specific sarcoma subtype
6. Prior Cancer Therapy . At least 3 weeks must have elapsed since the last cytotoxic chemotherapy or immunotherapy prior to leukapheresis/PBMC collection.

   * For targeted therapies, at least 4 half-lives or 3 weeks must have elapsed prior to leukapheresis (whichever is shorter).
7. Standard of care anti-cancer therapy will be permitted following leukapheresis but prior to initiation of cyclophosphamide such that:

   . At least 3 weeks must have elapsed since last cytotoxic chemotherapy or immunotherapy prior to starting treatment with cyclophosphamide.

   . For targeted therapies, at least 4 half-lives or 3 weeks must have elapsed prior to initiation of treatment with cyclophosphamide (whichever is shorter).

   . At least 2 weeks must have elapsed since last radiation therapy prior to cyclophosphamide.

   . Investigational anti-cancer therapy will not be permitted.
8. ECOG performance status of 0 or 1 (Performance level as measured by Karnofsky for patients . 16 years of age or Lansky for patients < 16 years of age, see Appendix B)
9. Participants must be willing to undergo tumor biopsy

   . Patients in whom biopsy is medically contraindicated or otherwise high risk will not be excluded and may forego research tumor biopsies
10. Patients must have organ and marrow function as defined below
11. Absolute neutrophil count (ANC) . 1 K/uL, Hemoglobin . 9 g/dL, Platelets.100 K/mm3
12. Serum creatinine . 2 mg/dL OR creatinine clearance > 50 mL/min
13. Aspartic transaminase (AST) . 1.5 x upper limit of normal (ULN), Alanine transaminase (ALT) . 1.5 x ULN, Bilirubin . 1.5 x ULN
14. Cardiac function . LVEF >50%
15. Pulmonary function

    . Oxygen saturation >92% on room air
    * Total lung capacity >70% of predicted
    * DLCO >60% of predicted
16. Women of childbearing potential (WOCBP) must agree to use method(s) of contraception: at least one highly effective or two effective accepted methods of contraception to avoid conception throughout the study in such a manner that the risk of pregnancy is minimized. Suggested precautions should be used to minimize the risk or pregnancy for at least 1 month before start of therapy, and while women are on study for up to 3 months after T cell infusion. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal
17. Men must be willing and able to use an acceptable method of birth control such as latex condom during the dosing period and for at least 3 months after completion of the study agent administration (T cell infusion) if their sexual partners are WOCBP.
18. Signed Informed Consent and if applicable, pediatric assent

Exclusion criteria:

1. Known sensitivity to cyclophosphamide and/or study agents Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener syndrome) within the past 2 years. Subjects with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
2. Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression. Subjects previously treated central nervous system metastases that are radiographically and neurologically stable for at least 6 weeks and do not require corticosteroids (of any dose) for symptomatic management for at least 14 days prior to first dose of attIL12-T cells are permitted to enroll. 3. Presence of metastatic disease in or near vital or critical structures that in the judgement of the treating physician in communication with PI or their delegate may lead to concern of immediate risk for harm from the inflammatory response.

4. Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment at the time of leukapheresis or attIL12 T cell infusion.

1. Standard of care anti-cancer therapy will be permitted following leukapheresis and prior to initiation of cyclophosphamide as bridging therapy (per section 12.4.1).
2. Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
3. In addition, local treatment (eg, by local surgery, radiotherapy, or ablation) of isolated lesions for palliative intent is acceptable beyond 30 days following attIL12 T cell administration with prior consultation and in agreement with the PI.
4. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5 Grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (eg, hearing loss) after consultation with the PI.
5. Investigational therapy for supportive care (e.g. COVID vaccine) will be permitted, as long as it is reviewed and discussed with the PI.

   5. History of primary immunodeficiency, solid organ transplantation, or previous clinical diagnosis of tuberculosis.

   6. Receipt of live, attenuated vaccine within 28 days prior to the first dose of investigational products 7. Major surgery (as defined by the investigator) within 4 weeks prior to first dose of treatment or if still recovering from prior surgery. Biopsy as per study protocol is allowed 8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs from the study agents, or compromise the ability of the subject to give written informed consent.

   9. Subjects with cognitive impairment, including adults with cognitive impairment such as trisomy 21 or similar conditions are not specifically excluded from participation, such that appropriate written informed consent is obtained from the parent or legal guardian and they are able to complete with the study protocol requirements and treatment.

   10. Active concurrent second malignancy 11. Pregnant or lactating women 12. Any positive test result for hepatitis B or C virus indicating acute or chronic infection 13. Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
To examine the incidence of adverse events. | through study completion; an average of 1 year.
  National Cancer Institute, Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. from screening through the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: John Livingston, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org